CLINICAL TRIAL: NCT03961516
Title: Glycemic Characterization and Pancreatic Imaging Correlates in Cystic Fibrosis
Acronym: CFCGM
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Katherine Kutney, Assistant Professor of Pediatric Endocrinology, University Hospitals Cleveland Medical Center
Other Study IDs: 20181150
Record Dates: First submitted 2019-05-16; First posted 2019-05-23 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis-related Diabetes; Cystic Fibrosis Liver Disease; Pancreatic Steatosis; Hepatic Steatosis
Keywords: continuous glucose monitor; cystic fibrosis; cystic fibrosis related diabetes
MeSH Terms: conditions — Cystic Fibrosis; Fatty Liver | interventions — Continuous Glucose Monitoring; Liver Extracts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Cystic Fibrosis, Pancreatic Sufficient: CF patients with exocrine pancreatic sufficiency
  Interventions: Device: Frequently Sampled Oral Glucose Tolerance Test and CGM; Radiation: MRI Pancreas and Liver
- Cystic Fibrosis, Pancreatic Insufficient, No Insulin: CF patients with exocrine pancreatic insufficiency but not treated with insulin therapy
  Interventions: Device: Frequently Sampled Oral Glucose Tolerance Test and CGM; Radiation: MRI Pancreas and Liver
- Cystic Fibrosis, Pancreatic Insufficient, Treated with Insulin: CF patients with exocrine pancreatic insufficiency who are treated with insulin therapy for CFRD
  Interventions: Device: Frequently Sampled Oral Glucose Tolerance Test and CGM; Radiation: MRI Pancreas and Liver

INTERVENTIONS:
Device: Frequently Sampled Oral Glucose Tolerance Test and CGM — Patients will undergo a 2 hour frequently sampled oral glucose tolerance test while wearing an active FreeStyle Libre Pro sensor. Using as a tool to collect data.
Radiation: MRI Pancreas and Liver — Patients will undergo an MRI of the pancreas and liver

SUMMARY:
The purpose of this study is to investigate the utility of a continuous glucose monitor device (CGM) in screening for cystic fibrosis related diabetes. The investigators will also study how fat deposition in the pancreas and liver impacts insulin production and response, as measured by a frequently sampled oral glucose tolerance test.

DETAILED DESCRIPTION:
Cystic Fibrosis Related Diabetes (CFRD) occurs in 20% of adolescents and 30-40% of adults with cystic fibrosis. CFRD is associated with reduced lung function, lower body mass index, and increased mortality. The CF Foundation recommends yearly Oral Glucose Tolerance Test (OGTT) for all CF patients beginning at age 10 years. Unfortunately adherence to screening recommendations is poor, with fewer than 50% of the eligible CF patients completing OGTT each year. Additionally, the OGTT has been criticized for poor reproducibility and for not accurately reflecting real-life glycemic excursions.

The FreeStyle Libre Pro is a blinded CGM that can record up to 14 days of home-living glucose data on one sensor. This quarter-sized device is placed on the upper arm and requires no fingerstick calibrations. Multiple studies have demonstrated the utility of CGM in CF patients, but no study has determined the utility of CGM in replicating the results of an OGTT. The use of CGM in CFRD screening has the potential to reduce screening burden, increase screening adherence and provide useful information about home glycemic excursions.

Pancreatic steatosis is common in CF with complete pancreatic fat replacement occurring in some cases. Pancreatic steatosis is also seen in patients with type 2 diabetes and may impact insulin secretion or the rate of beta cell decline. MRI is the most sensitive tool for detecting pancreatic steatosis. Ferrozzi described four patterns of pancreatic fat replacement in CF patients: (1) diffusely hyperintense with variable lobular pattern, (2) homogenous hyperintensity without lobular pattern, (3) hyperintense parenchyma with focal hypointensity, and (4) no structural or signal intensity changes. No studies have directly compared the degree of pancreatic steatosis with OGTT derived measures of insulin secretion or glycemic excursions on CGM.

Hepatic steatosis is also common in CF patients and has an unclear impact on insulin sensitivity. Outside of CF, hepatic steatosis is associated with insulin resistance.

This study has two aims:

Aim 1: Determine how closely the FreeStyle Libre Pro CGM can replicate the results of an in-clinic oral glucose tolerance test.

Aim 2: Explore whether pancreatic and hepatic steatosis correlated with insulin secretion and sensitivity in CF patients.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis confirmed by sweat chloride or genetics
* Pancreatic insufficient or pancreatic sufficient
* No change in insulin status (either initiating or discontinuing) in the past 3 months

Exclusion Criteria:

* CF liver disease with portal hypertension
* Systemic glucocorticoid exposure the past 2 weeks (does not include inhaled)
* Current pulmonary exacerbation treated with antibiotics
* Baseline or current FEV1 <30% at time of recruitment
* Transplant recipient
* Pancreatic sufficient on insulin
* Started CFTR modulator in the past 3 months

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with cystic fibrosis will be recruited from the LeRoy W. Matthews CF Center at UH Cleveland Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Glycemic agreement between plasma glucose and CGM | 0 min-120min
  Difference between blood glucose and CGM result will be calculated for each time point (0min, 30min, 60min, 90min, 120min).
Pancreatic Fat and Glycemic measures | 0min-120min
  Correlation between the degree of pancreatic fat replacement (Class 1-4 and fat fraction) and measures of beta cell function on glucose tolerance testing

SECONDARY OUTCOMES:
CGM results in CFRD vs. CFND | 0 min-120min
  Comparison of CGM parameters (time and excursions >140mg/dL and >200mg/dL between patients with insulin treated CFRD and no insulin treated CFRD
Pancreatic Fat by Modulator Status | 0min-120min
  Comparison of pancreatic fat (Ferrozzi category and fat fraction) in patients who are and are not receiving a CFTR modulator.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Kutney, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moran A, Dunitz J, Nathan B, Saeed A, Holme B, Thomas W. Cystic fibrosis-related diabetes: current trends in prevalence, incidence, and mortality. Diabetes Care. 2009 Sep;32(9):1626-31. doi: 10.2337/dc09-0586. Epub 2009 Jun 19. PMID 19542209
- [Background] Adler AI, Shine BS, Chamnan P, Haworth CS, Bilton D. Genetic determinants and epidemiology of cystic fibrosis-related diabetes: results from a British cohort of children and adults. Diabetes Care. 2008 Sep;31(9):1789-94. doi: 10.2337/dc08-0466. Epub 2008 Jun 5. PMID 18535191
- [Background] Annual Data Report 2016 Cystic Fibrosis Foundation Patient Registry [Internet]. Cystic Fibrosis Foundation Patient Registry. 2016
- [Background] Mainguy C, Bellon G, Delaup V, Ginoux T, Kassai-Koupai B, Mazur S, Rabilloud M, Remontet L, Reix P. Sensitivity and specificity of different methods for cystic fibrosis-related diabetes screening: is the oral glucose tolerance test still the standard? J Pediatr Endocrinol Metab. 2017 Jan 1;30(1):27-35. doi: 10.1515/jpem-2016-0184. PMID 27977404
- [Background] Walshaw M. Routine OGTT screening for CFRD - no thanks. J R Soc Med. 2009 Jul;102 Suppl 1(Suppl 1):40-4. doi: 10.1258/jrsm.2009.s19009. No abstract available. PMID 19605874
- [Background] Li A, Vigers T, Pyle L, Zemanick E, Nadeau K, Sagel SD, Chan CL. Continuous glucose monitoring in youth with cystic fibrosis treated with lumacaftor-ivacaftor. J Cyst Fibros. 2019 Jan;18(1):144-149. doi: 10.1016/j.jcf.2018.07.010. Epub 2018 Aug 10. PMID 30104123
- [Background] Leclercq A, Gauthier B, Rosner V, Weiss L, Moreau F, Constantinescu AA, Kessler R, Kessler L. Early assessment of glucose abnormalities during continuous glucose monitoring associated with lung function impairment in cystic fibrosis patients. J Cyst Fibros. 2014 Jul;13(4):478-84. doi: 10.1016/j.jcf.2013.11.005. Epub 2013 Dec 17. PMID 24359972
- [Background] Franzese A, Valerio G, Buono P, Spagnuolo MI, Sepe A, Mozzillo E, De Simone I, Raia V. Continuous glucose monitoring system in the screening of early glucose derangements in children and adolescents with cystic fibrosis. J Pediatr Endocrinol Metab. 2008 Feb;21(2):109-16. doi: 10.1515/jpem.2008.21.2.109. PMID 18422023
- [Background] O'Riordan SM, Hindmarsh P, Hill NR, Matthews DR, George S, Greally P, Canny G, Slattery D, Murphy N, Roche E, Costigan C, Hoey H. Validation of continuous glucose monitoring in children and adolescents with cystic fibrosis: a prospective cohort study. Diabetes Care. 2009 Jun;32(6):1020-2. doi: 10.2337/dc08-1925. Epub 2009 Mar 11. PMID 19279304
- [Background] Jefferies C, Solomon M, Perlman K, Sweezey N, Daneman D. Continuous glucose monitoring in adolescents with cystic fibrosis. J Pediatr. 2005 Sep;147(3):396-8. doi: 10.1016/j.jpeds.2005.05.004. PMID 16182684
- [Background] Della Corte C, Mosca A, Majo F, Lucidi V, Panera N, Giglioni E, Monti L, Stronati L, Alisi A, Nobili V. Nonalcoholic fatty pancreas disease and Nonalcoholic fatty liver disease: more than ectopic fat. Clin Endocrinol (Oxf). 2015 Nov;83(5):656-62. doi: 10.1111/cen.12862. Epub 2015 Aug 12. PMID 26201937
- [Background] Engjom T, Kavaliauskiene G, Tjora E, Erchinger F, Wathle G, Laerum BN, Njolstad PR, Frokjaer JB, Gilja OH, Dimcevski G, Haldorsen IS. Sonographic pancreas echogenicity in cystic fibrosis compared to exocrine pancreatic function and pancreas fat content at Dixon-MRI. PLoS One. 2018 Jul 26;13(7):e0201019. doi: 10.1371/journal.pone.0201019. eCollection 2018. PMID 30048483
- [Background] Ferrozzi F, Bova D, Campodonico F, De Chiara F, Uccelli M, Bacchini E, Grinzcich R, de Angelis GL, Battistini A. Cystic fibrosis: MR assessment of pancreatic damage. Radiology. 1996 Mar;198(3):875-9. doi: 10.1148/radiology.198.3.8628886.
- [Background] Lindblad A, Glaumann H, Strandvik B. Natural history of liver disease in cystic fibrosis. Hepatology. 1999 Nov;30(5):1151-8. doi: 10.1002/hep.510300527. PMID 10534335
- [Background] Ayoub F, Trillo-Alvarez C, Morelli G, Lascano J. Risk factors for hepatic steatosis in adults with cystic fibrosis: Similarities to non-alcoholic fatty liver disease. World J Hepatol. 2018 Jan 27;10(1):34-40. doi: 10.4254/wjh.v10.i1.34. PMID 29399276